CLINICAL TRIAL: NCT05469828
Title: Crizanlizumab Improves Tissue Oxygen Supply Demand Matching in Patients With Sickle Cell Anemia
Acronym: SEG101
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-21-00300
Record Dates: First submitted 2021-08-31; First posted 2022-07-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — crizanlizumab

STUDY DESIGN:
Intervention Model Description: Treatment and Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- treatment (Experimental): The effects of Crizanlizumab will be assessed in 20 nontransfused SCD subjects. After comprehensive baseline assessment one month prior the time of study initiation, patients will be started on 5mg/kg of body weight to be initiated at week 1 with follow up dosing at week 3 and week 7 then q4weeks until week 23, which will be the last dose given (7 total doses). Safety laboratories will be drawn at each infusion visit. There will be a follow up phone call the day after receiving the medication. Comprehensive blood and vascular testing will be repeated at Week 11 and Week 23 of treatment.
  Interventions: Drug: Crizanlizumab
- control (Active Comparator): A total of 10 SCD subjects will be recruited from the hematology clinic at CHLA, generating a similar distribution of SS and Sß0 hemoglobin. They will be studied twice, once at the beginning of the study, time 0, and once at the end of study, after 6 months. They will undergo the same cerebral, peripheral and cardiopulmonary testing procedures as the patients undergoing therapy. They will also have monthly phone calls to determine clinical outcomes such as crisis frequency, medication use, hospitalizations and other pertinent clinical findings that may arise.
  Interventions: Other: control

INTERVENTIONS:
Drug: Crizanlizumab — patients will be started on 5mg/kg of body weight to be initiated at week 1 with follow up dosing at week 3 and week 7 then q4weeks until week 23, which will be the last dose given (7 total doses).
  Arms: treatment
Other: control — Standard of care
  Arms: control

SUMMARY:
Hypothesis

Efficient unloading of oxygen to regions of high metabolic demand requires a healthy microvasculature to sense local oxygen tension and regulate flow, accordingly. In sickle cell disease patients, the investigators have demonstrated oxygen supply-demand mismatch, or SDM, in proportion to anemia severity. SDM occurs in both the peripheral circulation and the brain, and four characteristics: 1) Hyperemia beyond expected for the level of anemia, 2) Corresponding loss of vascular dilatory reserve, 3) Impaired oxygen unloading to the tissues, and 4) Tissue hypoxia. In sickle cell disease, red blood cell (RBC) and white blood cell (WBC) adhere to vascular endothelium triggering transient or irreversible microvascular damage as well as releasing vasoactive substances that contribute to microvascular dysregulation. The investigators postulate that ongoing microvascular damage/dysregulation in the setting of increased total blood flow contributes to SDM. The investigators believe SEG101, by lowering RBC and WBC adhesion to the microvasculature, will improve SDM and tissue oxygenation.

Objectives

* Primary - The investigators will test whether SEG101 improves SDM in patients with sickle cell anemia by measuring the change in tissue oxygenation measured by near infrared spectroscopy (NIRS).
* Secondary/Exploratory - The investigators will identify end-organ disease and whether improvement of SDM by SEG101 occurs in patients with sickle cell anemia.

DETAILED DESCRIPTION:
Objectives Primary Objectives 1. The investigators will test whether SEG101 improves Supply-Demand Matching in patients with sickle cell anemia measured by the change in tissue oxygenation by NIRS.

a) This is measured as a percent oxyhemoglobin saturation (%).

Secondary Objectives

1. Secondary measures to assess the change in tissue oxygenation will be

   1. In the somatic peripheral circulation - microcirculatory perfusion at rest and post-ischemia by laser doppler, venous oxygen saturation by venous blood gas and co-oximetry, and vasoconstriction by plethysmography.
   2. In the cerebral circulation - blood flow by arterial spin labeling, function brain MRI and response to CO2 challenge, sagittal sinus saturation by TRUST and tissue oxygen extraction by asymmetric spin echo.
   3. In the pulmonary vasculature - Pulmonary circulation - sleep study pulse oximetry for oxygenation and vasoconstriction by plethysmography, tricuspid regurgitant jet velocity (TRV) with echo markers of diastolic function to balance pulmonary vascular vs. left heart etiology of TRV.
2. Determine the relationship between SDM biomarkers and hemoglobin level (anemia).

   a) Hemoglobin and hematocrit for interaction between SDM and anemia
3. The investigators will determine whether low SDM predicts end-organ function in sickle cell anemia as compared to controls. These endpoints will be organ specific associations:

   a) eGFR and urinalysis for kidney, myocardial fibrosis, systolic/diastolic heart function, troponin and NT-pro-BNP
4. Relationship between markers of cellular adhesion, oxidative stress and inflammation, soluble VCAM and soluble P-selection.

   a) Interaction of SDM with soluble markers of adhesion and inflammation.
5. The investigators will identify interactions based on age and sex.

   a) Sex and gender related differences will act as covariates for all measures because many cardiovascular metrics have significant sex differences
6. Clinical Outcome Measures

   1. VOC history and prospective VOC burden.
   2. Blood pressure and ECG abnormalities/arrhythmias

Overall Design: The study will be performed at a single large sickle cell disease Centers of Excellence, Children's Hospital of Los Angeles in California, in 20 patients with sickle cell disease who will receive SEG101 therapy and 10 sickle cell anemia subjects who will not receive therapy. Full inclusion and exclusion criteria are defined in the human subjects section but sickle cell disease patients will be 16 years of age, or older (to be able to cooperate with the MRI examination without anesthesia), and free from hospitalization or emergency room visit for one month prior to the study. Entire cohort will be gender balanced.

The effects of SEG101 will be assessed in 20 nontransfused SCD subjects. Figure 3 summarizes the study schema. After comprehensive baseline assessment one month prior the time of study initiation, patients will be started on 5mg/kg of body weight to be initiated at week 1 with follow up dosing at week 3 and week 7 then q4weeks until week 23, which will be the last dose given (7 total doses). Safety laboratories will be drawn at each infusion visit. This will not be a randomized control trial. There will be a follow up phone call the day after receiving the medication. Comprehensive blood and vascular testing will be repeated at 3 and 6 months of treatment.

A total of 10 SCD subjects will be recruited from the hematology clinic at CHLA, generating a similar distribution of SS and Sß0 hemoglobin. The participants will be studied twice, once at the beginning of the study, time 0, and once at the end of study, after 6 months. The participants will undergo the same cerebral, peripheral and cardiopulmonary testing procedures as the patients undergoing therapy. The participants will also have monthly phone calls to determine clinical outcomes such as crisis frequency, medication use, hospitalizations and other pertinent clinical findings that may arise.

This is a non-randomized, open label intervention pilot study evaluating the effect of SEG101 on SDM in patients with sickle cell disease (SCD). The investigators plan to enroll 20 patients with SCD, who will receive SEG101. The investigators will also enroll 10 SCD subjects who will undergo all testing procedures but will not receive SEG101 treatment. The investigators will assess three vascular beds: 1. Peripheral circulation of the hand/arm (primary), 2. Brain (primary), and 3. Heart (exploratory).

Specific measures of SDM are summarized in Table 1. While SDM cannot currently be assessed in the heart, the heart represents a critical target for end organ dysfunction (Aim 2) because of its high metabolic demands and predisposition to microvascular damage.

Patient Population

Study Population - Patients with sickle cell anemia

Interruption or discontinuation of treatment

Patients may voluntarily withdraw from the study or be dropped from it at the discretion of the investigator at any time.

Treatment/Drug Administration

This is an open label study of SEG101. All patients will have peripheral SDM assessment in the arm/hand prior to and immediately following their initiation of SEG101 therapy. MRI exams will be performed prior to initiation of SEG101 therapy at the initial study visit but will not have immediate post therapy studies. Patients will have two repeat studies at 3-months and 6-months (end of study). The participants will receive SEG101 at 5mg/kg of body weight by intravenous infusion Qmonth and this will constitute "treatment".

Expected side effects

Previous research has demonstrated efficacy of SEG101 intravenous administration at 5mg/kg of body weight to decrease frequency of painful crisis. This is an FDA approved medication for prevention of painful crisis in SCD. In the Phase 2 clinical trial, the most common side effects noted were nausea (18%), arthralgia (18%), headache (17%), extremity pain (17%), back pain (15%), urinary tract infection (14%), musculoskeletal pain (12%), upper respiratory infection (11%), pyrexia (11%), diarrhea (11%), pruritis (8%), vomiting (8%), and chest pain (2%). These were derived from the SUSTAIN Phase 2 clinical trial.

Other medication use, standard of care

Standard of care therapies will not be stopped or changed. The investigators will encourage all practitioners to maintain pre-study medications throughout the study period, however, the investigators will not require it. The primary physician can adjust other medications as the participants determine necessary to their care. The SS patient's hydroxyurea use will be recorded in order to test a physiologic response (changes in brain and peripheral blood flow) and control for hydroxyurea effect. Use or non-use of hydroxyurea is not a contraindication to participating in this study, however, patients will need verbal assent from their primary hematologist to participate. HU therapy will need to be at the clinically tolerated dose for at least 6 months prior to starting the SEG101 therapy. HU therapy will not be adjusted or initiated during the study period and will not be considered a "treatment" for study purposes.

ELIGIBILITY:
Inclusion Criteria (Both Patient Groups - 1. SCD on SEG101 and 2. SCD not receiving SEG101)

* We will enroll only SS and Sß0 sickle cell disease patients
* Both male and female will be included.
* Our population of sickle cell disease is 90% African American and 10% Hispanic, therefore, our study population will reflect that distribution of ethnicity.
* Informed consent from legal guardian and/or patient
* Able to participate without needing sedation for MRI scan
* Age at least 16 years

Exclusion Criteria (Both Patient Groups - 1. SCD on SEG101 and 2. SCD not receiving SEG101)

* Any pain crisis requiring an ER visit and/or admission to the hospital and/or required parenteral pain medication in the previous 4 weeks.
* Any acute transfusion in the previous 4 weeks
* Need for chronic transfusion therapy
* Any known chronic illness that in the judgment of the investigator may compromise subject safety or data integrity. These include but are not limited to rheumatologic disorders, malignancy, severe asthma, chronic hepatic or renal insufficiency.
* Known pregnancy
* Seizure disorder
* Inability to cooperate with MRI examinations
* Contraindication to Crizanlizumab

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
The investigators will test whether SEG101 improves Supply-Demand Matching in patients with sickle cell anemia by measuring the change in tissue oxygenation by near infrared spectroscopy from baseline to 3 months and to 6 months. | Change measured over a 23 week period
  Tissue oxygenation is measured by near infrared spectroscopy in rSO2%. The investigators will account for changes in microcirculatory perfusion at rest and post-ischemia by laser doppler.

SECONDARY OUTCOMES:
The investigators will test whether SEG101 improves Supply-Demand Matching in patients with sickle cell anemia by measuring the change in microcirculatory perfusion at rest and post-ischemia | Change measured over a 23 week period
  Microcirculatory perfusion is measured by laser doppler in perfusion units (PU)
The investigators will test whether SEG101 improves Supply-Demand Matching in patients with sickle cell anemia by measuring the change in venous blood saturation and change in vessel endothelial function | Change measured over a 23 week period
  Venous oxygen saturation is measured by venous blood gas in pO2 and co-oximetry testing in percent saturation (% sat). Vasoconstriction is measured by plethysmography in percent change (% change).
The investigators will test whether SEG101 improves Supply-Demand Matching in patients with sickle cell anemia in the pulmonary vasculature using tricuspid regurgitant jet velocity as an estimate of pulmonary artery pressure. | Change measured over a 23 week period
  The tricuspid regurgitant jet velocity is a measure of pulmonary pressure and a predictor of mortality in sickle cell anemia measured in m/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Detterich, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] ITANO HA, PAULING L. A rapid diagnostic test for sickle cell anemia. Blood. 1949 Jan;4(1):66-8. No abstract available. PMID 18103217
- [Background] PAULING L, ITANO HA, et al. Sickle cell anemia a molecular disease. Science. 1949 Nov 25;110(2865):543-8. doi: 10.1126/science.110.2865.543. No abstract available. PMID 15395398
- [Background] Chien S, Usami S, Bertles JF. Abnormal rheology of oxygenated blood in sickle cell anemia. J Clin Invest. 1970 Apr;49(4):623-34. doi: 10.1172/JCI106273. PMID 5443167
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Steiner CA, Miller JL. Sickle Cell Disease Patients in U.S. Hospitals, 2004. 2006 Dec. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #21. Available from http://www.ncbi.nlm.nih.gov/books/NBK63489/ PMID 21938835
- [Background] Niss O, Fleck R, Makue F, Alsaied T, Desai P, Towbin JA, Malik P, Taylor MD, Quinn CT. Association between diffuse myocardial fibrosis and diastolic dysfunction in sickle cell anemia. Blood. 2017 Jul 13;130(2):205-213. doi: 10.1182/blood-2017-02-767624. Epub 2017 May 15. PMID 28507082
- [Background] Kato GJ, Gladwin MT, Steinberg MH. Deconstructing sickle cell disease: reappraisal of the role of hemolysis in the development of clinical subphenotypes. Blood Rev. 2007 Jan;21(1):37-47. doi: 10.1016/j.blre.2006.07.001. Epub 2006 Nov 7. PMID 17084951
- [Background] Detterich JA, Kato RM, Rabai M, Meiselman HJ, Coates TD, Wood JC. Chronic transfusion therapy improves but does not normalize systemic and pulmonary vasculopathy in sickle cell disease. Blood. 2015 Aug 6;126(6):703-10. doi: 10.1182/blood-2014-12-614370. Epub 2015 Jun 2. PMID 26036801
- [Background] Friedman D, Szmuszkovicz J, Rabai M, Detterich JA, Menteer J, Wood JC. Systemic endothelial dysfunction in children with idiopathic pulmonary arterial hypertension correlates with disease severity. J Heart Lung Transplant. 2012 Jun;31(6):642-7. doi: 10.1016/j.healun.2012.02.020. Epub 2012 Mar 21. PMID 22440720
- [Background] Kato GJ, Hebbel RP, Steinberg MH, Gladwin MT. Vasculopathy in sickle cell disease: Biology, pathophysiology, genetics, translational medicine, and new research directions. Am J Hematol. 2009 Sep;84(9):618-25. doi: 10.1002/ajh.21475. PMID 19610078
- [Background] Delpy DT, Cope MC, Cady EB, Wyatt JS, Hamilton PA, Hope PL, Wray S, Reynolds EO. Cerebral monitoring in newborn infants by magnetic resonance and near infrared spectroscopy. Scand J Clin Lab Invest Suppl. 1987;188:9-17. PMID 2835812
- [Background] Tenland T, Salerud EG, Nilsson GE, Oberg PA. Spatial and temporal variations in human skin blood flow. Int J Microcirc Clin Exp. 1983;2(2):81-90. PMID 6236158
- [Background] Thorniley MS, Houston R, Wickramasinghe YA, Rolfe P. Application of near-infrared spectroscopy for the assessment of the oxygenation level of myoglobin and haemoglobin in cardiac muscle in vivo. Biochem Soc Trans. 1990 Dec;18(6):1195-6. doi: 10.1042/bst0181195. No abstract available. PMID 2088860
- [Background] Nilsson GE, Tenland T, Oberg PA. Evaluation of a laser Doppler flowmeter for measurement of tissue blood flow. IEEE Trans Biomed Eng. 1980 Oct;27(10):597-604. doi: 10.1109/TBME.1980.326582. No abstract available. PMID 6449469
- [Background] Lee JH, Jang YE, Song IK, Kim EH, Kim HS, Kim JT. Near-Infrared Spectroscopy and Vascular Occlusion Test for Predicting Clinical Outcome in Pediatric Cardiac Patients: A Prospective Observational Study. Pediatr Crit Care Med. 2018 Jan;19(1):32-39. doi: 10.1097/PCC.0000000000001386. PMID 29140967
- [Background] De Blasi RA, Cope M, Ferrari M. Oxygen consumption of human skeletal muscle by near infrared spectroscopy during tourniquet-induced ischemia in maximal voluntary contraction. Adv Exp Med Biol. 1992;317:771-7. doi: 10.1007/978-1-4615-3428-0_94. No abstract available. PMID 1288203
- [Background] Adams RJ, McKie VC, Brambilla D, Carl E, Gallagher D, Nichols FT, Roach S, Abboud M, Berman B, Driscoll C, Files B, Hsu L, Hurlet A, Miller S, Olivieri N, Pegelow C, Scher C, Vichinsky E, Wang W, Woods G, Kutlar A, Wright E, Hagner S, Tighe F, Waclawiw MA, et al. Stroke prevention trial in sickle cell anemia. Control Clin Trials. 1998 Feb;19(1):110-29. doi: 10.1016/s0197-2456(97)00099-8. PMID 9492971
- [Background] Adams RJ, McKie VC, Hsu L, Files B, Vichinsky E, Pegelow C, Abboud M, Gallagher D, Kutlar A, Nichols FT, Bonds DR, Brambilla D. Prevention of a first stroke by transfusions in children with sickle cell anemia and abnormal results on transcranial Doppler ultrasonography. N Engl J Med. 1998 Jul 2;339(1):5-11. doi: 10.1056/NEJM199807023390102. PMID 9647873
- [Background] Nathan DG. Regulation of fetal hemoglobin synthesis by cell cycle specific drugs. Prog Clin Biol Res. 1985;191:475-500. No abstract available. PMID 2413483
- [Background] Gordeuk VR, Castro OL, Machado RF. Pathophysiology and treatment of pulmonary hypertension in sickle cell disease. Blood. 2016 Feb 18;127(7):820-8. doi: 10.1182/blood-2015-08-618561. Epub 2016 Jan 12. PMID 26758918
- [Background] Presley TD, Perlegas AS, Bain LE, Ballas SK, Nichols JS, Sabio H, Gladwin MT, Kato GJ, Kim-Shapiro DB. Effects of a single sickling event on the mechanical fragility of sickle cell trait erythrocytes. Hemoglobin. 2010;34(1):24-36. doi: 10.3109/03630260903546999. PMID 20113285
- [Background] Reiter CD, Wang X, Tanus-Santos JE, Hogg N, Cannon RO 3rd, Schechter AN, Gladwin MT. Cell-free hemoglobin limits nitric oxide bioavailability in sickle-cell disease. Nat Med. 2002 Dec;8(12):1383-9. doi: 10.1038/nm1202-799. Epub 2002 Nov 11. PMID 12426562